CLINICAL TRIAL: NCT05093023
Title: ABCB1 Single Nucleotide Polymorphism Genotypes as Predictors of Paclitaxel-Induced Peripheral Neuropathy in Breast Cancer
Brief Title: ABCB1 SNPs as Predictors of PIPN
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, nabil mahmoud, Master's Student, Ain Shams University
Other Study IDs: ABCB1 in Paclitaxel Neuropathy
Record Dates: First submitted 2021-10-13; First posted 2021-10-26 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Paclitaxel Adverse Reaction; Neuropathy;Peripheral; Breast Cancer
MeSH Terms: conditions — Neuritis; Breast Neoplasms | interventions — Real-Time Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: Real-Time PCR — Genomic DNA was extracted from 2 ml of venous blood. ABCB1 1236 G>A and 3435 G>A were genotyped using predesigned TaqMan SNP genotyping assays on a stepOne PCR instrument in accordance with the manufacturer's protocol.

SUMMARY:
The study aim is to determine the allele frequencies of 1236 G>A and 3435 G>A in ABCB1 and study their association with the incidence and severity of paclitaxel-induced peripheral neuropathy while adjusting for other baseline covariates in Egyptian patients. Additionally, the study aimed at fitting and validating logistic regression models with the aforementioned SNPs evaluated in additive, dominant, overdominant, and recessive genetic models and performing diagnostics for the best model in terms of internal validity.

ELIGIBILITY:
Inclusion Criteria:

1. Egyptian females ≥18 years of age.
2. Histologically confirmed Breast Cancer.
3. Receiving conventional neoadjuvant or adjuvant weekly paclitaxel.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
5. Adequate organ reserves ((serum creatinine ≤1.5x upper normal limit (UNL), total bilirubin ≤1.5x UNL, absolute neutrophil count ≥1.5 x 10^9/L, platelet count ≥100 x 10^9/L, AST and ALT ≤3.0x UNL, and alkaline phosphatase ≤3.0x UNL).
6. No major neurological disease or symptoms prior to the start of paclitaxel therapy.
7. neither subjective nor objective evidence of metastatic disease.

Exclusion Criteria:

1. Pregnancy.
2. Patients with recurrent or metastatic (local or distant) breast cancer.
3. Neuropathic at the time of recruitment.
4. History of neuropathy prior to recruitment.
5. Previously exposed to taxanes or any other microtubule Inhibitors, or regimens including platinates.
6. Patients currently receiving dose-dense biweekly taxane-containing regimens.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Egyptian women with histologically confirmed Breast Cancer, receiving neoadjuvant and/or adjuvant weekly paclitaxel-containing regimens.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Grade 2 or higher peripheral neuropathy | 12 weeks
  Grade 2 or higher peripheral neuropathy evaluated by the National Cancer Institute Common Toxicity Criteria (version 5.0)

CONTACTS AND LOCATIONS:
Locations (1):
- Nasser's Institute Hospital, Cairo, Aghakhan, Egypt

REFERENCES:
- [Background] Green H, Soderkvist P, Rosenberg P, Mirghani RA, Rymark P, Lundqvist EA, Peterson C. Pharmacogenetic studies of Paclitaxel in the treatment of ovarian cancer. Basic Clin Pharmacol Toxicol. 2009 Feb;104(2):130-7. doi: 10.1111/j.1742-7843.2008.00351.x. Epub 2008 Dec 16. PMID 19143748
- [Background] Kimchi-Sarfaty C, Marple AH, Shinar S, Kimchi AM, Scavo D, Roma MI, Kim IW, Jones A, Arora M, Gribar J, Gurwitz D, Gottesman MM. Ethnicity-related polymorphisms and haplotypes in the human ABCB1 gene. Pharmacogenomics. 2007 Jan;8(1):29-39. doi: 10.2217/14622416.8.1.29. PMID 17187507
- [Background] Rivera E, Cianfrocca M. Overview of neuropathy associated with taxanes for the treatment of metastatic breast cancer. Cancer Chemother Pharmacol. 2015 Apr;75(4):659-70. doi: 10.1007/s00280-014-2607-5. Epub 2015 Jan 18. PMID 25596818
- [Background] Scripture CD, Figg WD, Sparreboom A. Peripheral neuropathy induced by paclitaxel: recent insights and future perspectives. Curr Neuropharmacol. 2006 Apr;4(2):165-72. doi: 10.2174/157015906776359568. PMID 18615126
- [Background] Gao B, Russell A, Beesley J, Chen XQ, Healey S, Henderson M, Wong M, Emmanuel C, Galletta L, Johnatty SE, Bowtell D; Australian Ovarian Cancer Study Group; Haber M, Norris M, Harnett P, Chenevix-Trench G, Balleine RL, deFazio A. Paclitaxel sensitivity in relation to ABCB1 expression, efflux and single nucleotide polymorphisms in ovarian cancer. Sci Rep. 2014 May 9;4:4669. doi: 10.1038/srep04669. PMID 24810093
- [Background] Sparreboom A, van Tellingen O, Nooijen WJ, Beijnen JH. Preclinical pharmacokinetics of paclitaxel and docetaxel. Anticancer Drugs. 1998 Jan;9(1):1-17. doi: 10.1097/00001813-199801000-00001. PMID 9491787
- [Background] Wolking S, Schaeffeler E, Lerche H, Schwab M, Nies AT. Impact of Genetic Polymorphisms of ABCB1 (MDR1, P-Glycoprotein) on Drug Disposition and Potential Clinical Implications: Update of the Literature. Clin Pharmacokinet. 2015 Jul;54(7):709-35. doi: 10.1007/s40262-015-0267-1. PMID 25860377
- [Background] Tulsyan S, Mittal RD, Mittal B. The effect of ABCB1 polymorphisms on the outcome of breast cancer treatment. Pharmgenomics Pers Med. 2016 Apr 27;9:47-58. doi: 10.2147/PGPM.S86672. eCollection 2016. PMID 27175090
- [Background] Cavaletti G, Marmiroli P. Chemotherapy-induced peripheral neurotoxicity. Nat Rev Neurol. 2010 Dec;6(12):657-66. doi: 10.1038/nrneurol.2010.160. Epub 2010 Nov 9. PMID 21060341